CLINICAL TRIAL: NCT03221205
Title: Effect of Nasal CPAP on Myocardial Dysfunction and Glycemic Control in Patients With Type 2 Diabetes, Obstructive Sleep Apnea and Obesity
Brief Title: Effect of CPAP on Myocardial Dysfunction in Type 2 Diabetes Mellitus and Obstructive Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Collaborators: Fundación Clínica Médica Sur (Other); National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Armando Castorena-Maldonado, Head of Otolaryngology Department, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C_30-13
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2; Continuous Positive Airway Pressure; Myocardial Dysfunction; Echocardiography; Obesity
Keywords: sleep apnea, obstructive; obesity; DM2; TEI index; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham CPAP (Sham Comparator): Patients randomized to use sham CPAP via a nasal mask every night for three months, also with medical treatment for control of obesity, optimal medical treatment for diabetes mellitus.
  Interventions: Device: Sham CPAP
- Therapeutic CPAP (Experimental): Patients randomized to use CPAP programmed to administer automatically pressure from 4 to 20 cm H2O via a nasal mask every night for three months, also with medical treatment for control of obesity, optimal medical treatment for diabetes mellitus.
  Interventions: Device: Therapeutic CPAP

INTERVENTIONS:
Device: Sham CPAP — CPAP (ResMed AutoSet S9 with humidifier) to be used by the participant via nasal mask and tube, programmed to apply 0.5 cmH2O (measured at the nasal mask) via a resistance to assure the lack of distal pressure.
  Arms: Sham CPAP
Device: Therapeutic CPAP — Use of CPAP (ResMed AutoSet S9 with humidifier) through nasal mask and tube with automatized pressure from 4 to 20 cmH2O.
  Arms: Therapeutic CPAP

SUMMARY:
This study evaluates the effect of the use of nasal CPAP in the cardiac function, measured by strain and TEI index, in patients with type 2 diabetes mellitus, obstructive sleep apnea and obesity. In order to do so, 76 patients will be studied, half will use sham CPAP and half will use therapeutic CPAP for three months, with echocardiogram, laboratory studies, ambulatory monitoring of arterial tension and sleep study before and after CPAP use.

DETAILED DESCRIPTION:
The obstructive sleep apnea syndrome (OSAS) is a disease characterized by repeated episodes of partial of total obstruction of the upper airway during sleep. It affects 3.2% of adults in Mexico City. These patients have a higher risk of suffering traffic accidents, cardiovascular diseases, a lower quality of life and premature death. The association between OSAS and heart failure is complex, but it is known that they have a higher risk of myocardial dysfunction with OR 2.4 (IC 95% 1.2 - 4.6), with higher mortality against controls. Type 2 diabetes mellitus (DM2) is a chronic metabolic disease that leads to macro and micro vascular damage, and is the first cause of mortality in Mexico (13.8% of all deaths in people older than 20 years). Its general prevalence in adults is of 7%. There is a strong association between OSAS, insulin resistance and DM2, with studies with 86% of patients with DM2 having some degree of sleep apnea reported, with 22.6% having severe OSAS. The presence of DM2 doubles the risk of cardiovascular disease in men and triples it in women, with coronary cardiac disease being the main cause of death. Patients with OSAS have altered myocardial function even in asymptomatic state, also patients with DM2 have been shown to have abnormalities in myocardial function, myocardial performance and myocardial elongation in comparison with a control group. There is no current information about the effect of treatment with CPAP on myocardial performance of patients with OSAS, DM2 and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical data of obstructive sleep apnea: snoring, witnessed apneas, excessive daytime somnolence.
* Previous diagnosis of type 2 diabetes mellitus, with medical treatment according to the ADA 2012 guidelines, but only with one of the next drugs: biguanides, sulphonylurea, meglitinide, thiazolidinedione, alpha-glucosidase inhibitors.
* Obesity, defined by a body mass index higher than 29 kilogram per square meter.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Insulin dependent type 2 diabetes mellitus
* Fasting plasma glucose higher than 212 mg/dL .
* Antecedent of myocardial infarction, heart failure or arrhythmia.
* Obstructive sleep apnea in treatment.
* Urgent need of CPAP treatment (public transport drivers, heavy machine operators).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
TEI index | After 3 months of CPAP use.
  Cardiac performance, evaluated through TEI index.
Strain | After 3 months of CPAP use.
  Cardiac performance, evaluated through echocardiographic strain.

SECONDARY OUTCOMES:
Hemoglobin A1C | After three months of CPAP use.
  Glycemic control via hemoglobin A1C, percent.
Plasma glucose. | After 3 months of CPAP use.
  Levels of glucose in plasma, in mg/dL.
Apnea hypopnea index | After 3 months CPAP use.
  Number of events of apnea and hypopnea per hour of sleep, evaluated through an type 3 overnight sleep study,
Mean oxygen saturation | After 3 months of CPAP use.
  Mean value of the data of oxygen saturation reported in a type 3 overnight sleep study.
Time of hypercapnia | After 3 months of CPAP use.
  Number of minutes per night of sleep in which the carbon dioxide value was above 45 mmHg, as measured via transcutaneous capnography in an overnight sleep study.
Time of hypercapnia | After three months CPAP use.
  Number of minutes per night of sleep in which the carbon dioxide value was above 45 mmHg, as measured via transcutaneous capnography in an overnight sleep study.
Mean CO2 | After three months CPAP use
  Mean of the values of carbon dioxide during a night of sleep, as measured via transcutaneous capnography in an overnight sleep study.
Highest CO2 | After three months CPAP use
  Highest reported value of carbon dioxide during a night of sleep, as measured via transcutaneous capnography in an overnight sleep study.
Time of saturation under 90%. | After 3 months CPAP use
  Percent of the time of duration of a type three overnight sleep study in which the SO2 was under 90%.
Mean value of arterial pressure | After 3 months of CPAP use
  Mean value of systolic and diastolic arterial pressure, as measured through an ambulatory monitoring of arterial pressure for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Armando R Castorena-Maldonado, MD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Insituto Nacional de Enfermedades Respiratorias, Mexico City, Delegacion Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ernande L, Rietzschel ER, Bergerot C, De Buyzere ML, Schnell F, Groisne L, Ovize M, Croisille P, Moulin P, Gillebert TC, Derumeaux G. Impaired myocardial radial function in asymptomatic patients with type 2 diabetes mellitus: a speckle-tracking imaging study. J Am Soc Echocardiogr. 2010 Dec;23(12):1266-72. doi: 10.1016/j.echo.2010.09.007. Epub 2010 Oct 8. PMID 20932716
- [Background] Ng AC, Delgado V, Bertini M, van der Meer RW, Rijzewijk LJ, Shanks M, Nucifora G, Smit JW, Diamant M, Romijn JA, de Roos A, Leung DY, Lamb HJ, Bax JJ. Findings from left ventricular strain and strain rate imaging in asymptomatic patients with type 2 diabetes mellitus. Am J Cardiol. 2009 Nov 15;104(10):1398-401. doi: 10.1016/j.amjcard.2009.06.063. Epub 2009 Sep 26. PMID 19892057
- [Background] Marwick TH. Tissue Doppler imaging for evaluation of myocardial function in patients with diabetes mellitus. Curr Opin Cardiol. 2004 Sep;19(5):442-6. doi: 10.1097/01.hco.0000131535.32657.87. PMID 15316450
- [Background] Carrillo-Alduenda JL, Arredondo del Bosque F, Reyes-Zúñiga M, Barabia Ortega B, Yáñez-Gutiérrez L, Torre-Bouscoulet L, Castorena-Maldonado A. Índice de funcionamiento miocárdico en pacientes con síndrome de apnea obstructiva del sueño. Neumología y cirugía de tórax. 2009;68(3):100-105
- [Background] Tugcu A, Yildirimturk O, Tayyareci Y, Demiroglu C, Aytekin S. Evaluation of subclinical right ventricular dysfunction in obstructive sleep apnea patients using velocity vector imaging. Circ J. 2010 Feb;74(2):312-9. doi: 10.1253/circj.cj-09-0562. Epub 2009 Dec 15. PMID 20009388